CLINICAL TRIAL: NCT06277206
Title: A Study Using 18F-FAPI PET to Evaluate Pathologic Response to Systemic Treatment in Pancreatic Adenocarcinoma
Brief Title: A Study Using 18F-FAPI PET to Evaluate Treatment Response in Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Other Study IDs: FAPIPDAC02
Record Dates: First submitted 2024-02-17; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: 18F-FAPI; Pancreas Adenocarcinoma; Systemic Treatment; Pathologic Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-FAPI PET/CT — Enrolled patients underwent 18F-FAPI PET/CT at diagnosis. And preoperative 18F-FAPI PET/CT was completed in the patients met the criteria for conversion surgery after systemic treatment. The correlation between changes of parameters before and after treatment and pathologic response was analyzed.

SUMMARY:
To explore the potential utility of 18F-FAPI-04 PET/CT for pathologic response evaluation to systemic treatment in PDAC

ELIGIBILITY:
Inclusion Criteria:

* suspected to have pancreatic cancer by radiological imaging
* planned systemic treatment
* possibility of conversion surgery
* willingness to participate the study

Exclusion Criteria:

* without pathologically confirmed pancreatic cancer
* poor performance status or organ functions that cannot meet the systemic treatment requirements
* metastatic disease
* pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients with resectable, borderline or locally advanced disease who plan to undergo systemic treatment, including chemotherpy or chemoimmunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Change of Maximum standardized uptake value | Baseline and preoperation
  Change of SUVmax before and after treatment
Change of Mean standardized uptake value | Baseline and preoperation
  Change of SUVmean before and after treatment

SECONDARY OUTCOMES:
Maximum standardized uptake value | Baseline
  Baseline SUVmax at diagnosis
Mean standardized uptake value | Baseline
  Baseline SUVmean at diagnosis
Metabolic Tumor Volume | Baseline
  Baseline MTV at diagnosis
Total Lesion FAP expression | Baseline
  Baseline TLF at diagnosis
Change of Metabolic Tumor Volume | Baseline and preoperation
  Change of MTV before and after treatment
Change of Total Lesion FAP expression | Baseline and preoperation
  Change of TLF before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No